CLINICAL TRIAL: NCT01593488
Title: Multicentered Phase II Study Evaluating the Activity and Toxicity of Liposomal Cytarabine in the Treatment of Children and Adolescents With Acute Lymphoblastic Leukemia With Resistent or Relapsed Central Nervous System Involvement
Brief Title: Liposomal Cytarabine in the Treatment of Central Nervous System Resistant or Relapsed Acute Lymphoblastic Leukemia in Children
Acronym: CILI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Collaborators: Santobono-Pausilpon Hospital (Unknown); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); University of Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CILI; 2011-002622-48 (EudraCT Number)
Record Dates: First submitted 2012-04-27; First posted 2012-05-08 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: recurrent; CNS disease; intrathecal therapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence; Central Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intrathecal liposomal cytarabine (Experimental)
  Interventions: Drug: liposomal cytarabine

INTERVENTIONS:
Drug: liposomal cytarabine — given intrathecally in induction phase every 15 days until CSF response for up to 7 injections. Then it is given every 4 weeks during consolidation phase while patient awaiting bone marrow transplant. For those patients who are not candidates for a bone marrow transplant, the drug will be given every 3 months for 4 administrations (maintenance therapy)

SUMMARY:
The purpose of this study is to describe the activity and toxicity of a new formulation of cytarabine called liposomal cytarabine given into the central nervous system for the treatment of central nervous system localization of acute lymphoblastic leukemia (ALL) in children and adolescents.

DETAILED DESCRIPTION:
Liposomal cytarabine (DepoCyte) is a new formulation of the drug cytarabine, a drug commonly used in the treatment of ALL. This formulation of the drug can be given intrathecally (into the spinal fluid), and is released slowly over a longer period, about two weeks. This allows a longer exposure of the drug to the central nervous system, and requires fewer intrathecal injections for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years
* Diagnosis of acute lymphoblastic leukemia (ALL)
* Central nervous system involvement with malignant cells present in cerebrospinal fluid
* CNS involvement may be refractive to prior systemic therapy, a first recurrence after prior systemic and intrathecal therapy or a second recurrence
* CNS involvement may be an isolated lesion or present with other sites of disease
* ECOG performance status 0-2
* Life expectancy of at least 8 weeks
* Absence of severe organ dysfunction
* Informed consent

Exclusion Criteria:

* Eligibility for AIEOP studies of first recurrence of ALL,and receiving therapy in a center participating in the AIEOP studies
* Concurrent treatment with experimental therapies
* Severe neurologic toxicities from previous chemotherapy
* Severe coagulopathy at time of recurrence
* Sepsis
* Intrathecal therapy within 1 week of planned study therapy
* Total body or head and spine radiation within 8 weeks of enrolment
* Bone marrow transplant within 8 weeks of start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2012-03; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
number of cerebrospinal fluid (CSF) responses | from two weeks after date of patient registration until the date of second consecutive cerebrospinal fluid exam that is negative for malignant cells, up to 12 weeks
number of patients with grade 3 or higher neurological adverse events, excluding headache) according to CTCAE 4.02 | assessed from date of patient registration to date of cerebrospinal fluid response, up to 12 weeks

SECONDARY OUTCOMES:
time to reaching CSF response | date of patient registration to date of CSF response, up to 12 weeks
  date of reaching CSF response is the first date of two consecutive negative cytomorphologic exams of CSF
duration of CSF response | up to 12 months
  duration of response is the length of time in days from the date of the CSF response to the date of the first positive cytomorphologic CSF exam
worst grade non neurologic Adverse event during induction, according to CTCAE 4.02 | up to 12 weeks
worst grade toxicity after induction therapy according to CTCAE 4.02 | up to 12 months
  Measured from date of CSF response
overall survival | one year
time from patient registration to progression of disease in non CNS site | up to one year
concentration of study drug present in CSF at each induction therapy | prior to each induction therapy at 15 day intervals for up to 6 cycles
correlation of activity and toxicity with residual study drug level in CSF during induction | measured at 15 day intervals for up to 6 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Rosanna Parasole, M.D., Principal Investigator — Santobono-Pausilipon Hospital; Massimo Di Maio, M.D., Principal Investigator — National Cancer Institute, Naples; Francesco Perrone, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; A. Pession, Principal Investigator — Policlinico S. Orsola-Malpighi, Bologna; William Morello, Principal Investigator — Policlinico S. Orsola-Malpighi, Bologna; E. Strocchi, Principal Investigator — University of Bologna
Locations (10):
- Italy (10):
  - P.O. Gaspare Rodolico, Catania
  - Istituto G. Gasilini, Genova
  - Ospedale S. Gerardo Clinica Pediatrica, Monza
  - AORN Santobon - Pauslipon, Napoli
  - A.O. Università Padova, Padua
  - ARNAS Osp Civico di Cristina, Palermo
  - IRCCS Ospedale Bambino Gesu', Roma
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - IRCCS Burlo Garofalo Istituto per l'Infanzia Emato Oncologia, Trieste
  - Ospedale Policlinico G.B. Rossi, Verona